CLINICAL TRIAL: NCT05755282
Title: Touch and Feel Evaluation of Two Foam Hand Sanitizers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MED-2022-DIV60-001
Record Dates: First submitted 2023-02-03; First posted 2023-03-06 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hand Hygiene
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants will try all products. Participants are randomized to the order of study product application.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A: spectrum first then Purell (Active Comparator): Half of participants will apply Spectrum Advanced (#1) Hand Sanitizer Foam followed by Purell Advanced (#2) Hand Sanitizer Foam
  Interventions: Drug: Post-market foam alcohol-based hand sanitizer #1; Drug: Post-market foam alcohol-based hand sanitizer #2
- B: Purell first then spectrum (Active Comparator): Half of participants will apply hand Purell Advanced (#2) Hand Sanitizer Foam followed by Spectrum Advanced (#1) Hand Sanitizer
  Interventions: Drug: Post-market foam alcohol-based hand sanitizer #1; Drug: Post-market foam alcohol-based hand sanitizer #2

INTERVENTIONS:
Drug: Post-market foam alcohol-based hand sanitizer #1 — Automated dispenser will dispense 1 mL of hand sanitizer product onto hands.
  Other Names: Spectrum™ Advanced Hand Sanitizer Foam #1
Drug: Post-market foam alcohol-based hand sanitizer #2 — Automated dispenser will dispense 1 mL of hand sanitizer product onto hands.
  Other Names: PURELL® Advanced Foam Hand sanitizer #2

SUMMARY:
Hand sanitizers are a standard of hygiene requirements. Hand sanitizers must be effective at reducing germ count on the hands while ideally providing emollients to moisturize the skin after use. To improve compliance with hand sanitizing protocols, hand sanitizers should provide a pleasant touch and feel experience for end users, especially for healthcare worker (HCW) users, who use these products frequently.

DETAILED DESCRIPTION:
Hand sanitizers are a standard of hygiene requirements. Hand sanitizers are a standard tool frequently used in hospital settings by healthcare (HCWs) for hand disinfection. The Centers for Disease Control and Prevention (CDC) states that HCWs should use an alcohol-based hand rub, such as a hand sanitizer, or wash their hands with soap and water immediately before and after patient contact, during aseptic tasks, after contact with blood, bodily fluids, or contaminated surfaces, and immediately after glove removal. 1 Additionally, the World Health Organization (WHO) guidelines on hand hygiene state that alcohol-based handrubs rapidly and effectively inactivate a wide array of potentially harmful microorganisms on hands. 2 Hand sanitizers must be effective at reducing germ count on the hands while ideally providing emollients to moisturize the skin after use. To improve compliance with hand sanitizing protocols, hand sanitizers should provide a pleasant touch and feel experience for users, especially for healthcare worker (HCW) users.

The goal of this study is to evaluate the user touch and feel experience of two hand sanitizer foam products produced by Medline and GOJO when the products are used by HCWs.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers ≥ 18 years of age

Exclusion Criteria:

* Individual has a skin condition that might result in irritation from the hand sanitizers.
* Individual has a known allergy to the ingredients in the test products.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyce JM, Pittet D; Healthcare Infection Control Practices Advisory Committee; HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Guideline for Hand Hygiene in Health-Care Settings. Recommendations of the Healthcare Infection Control Practices Advisory Committee and the HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Society for Healthcare Epidemiology of America/Association for Professionals in Infection Control/Infectious Diseases Society of America. MMWR Recomm Rep. 2002 Oct 25;51(RR-16):1-45, quiz CE1-4. PMID 12418624
- [Background] WHO Guidelines on Hand Hygiene in Health Care: First Global Patient Safety Challenge Clean Care Is Safer Care. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK144013/ PMID 23805438

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants sampled both products (Spectrum and Purell). The order in which they sampled the products was randomized according to a randomization table.
Groups:
- Arm A: Spectrum First Than Purell: Arm A participants first applied spectrum hand sanitizer followed by a washout period. They then applied Purell hand sanitizer.
- Arm B: Purell First Than Spectrum: Arm B participants first applied purell hand sanitizer followed by a washout period. They then applied spectrum hand sanitizer.
Period: Overall Study
Arm/Group | Arm A: Spectrum First Than Purell | Arm B: Purell First Than Spectrum
Started | 19 | 27
Completed | 19 | 26
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants were randomized using a randomization table to either Arm A or Arm B
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Spectrum First Than Purell | Arm B: Purell First Than Spectrum | Total
Number analyzed (Participants) | 19 | 26 | 45
Age, Continuous [Mean (Full Range); unit: years] — participants were asked to report their age.
  years
    Age by Arm | 42.63 [26 to 63] | 42.00 [21 to 62] | 42.27 [21 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective Foam Sanitizer User Touch and Feel Experience
Description: The user touch and feel experience of the foam hand sanitizer products evaluated by visual analog scale assessments (VAS) ranging from 0 to 100, with higher scores indicating a more favorable outcome, of healthcare workers overall satisfaction and moisturization.
Time Frame: up to 30 mins to complete on a single day; Directly after participants hands have dried after application of each hand sanitizer product
Population: Participants were asked to answer four questions about each of the products and then asked which product they preferred (see preference outcome measure documented separately)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm A Spectrum Frist Than Purell: Arm A participants first applied spectrum hand sanitizer followed by a washout period, then applied purell hand sanitizer.
- Arm B Purell First Than Spectrum: Arm B participants first applied purell hand sanitizer followed by a washout period, then applied spectrum hand sanitizer.
Arm/Group | Arm A Spectrum Frist Than Purell | Arm B Purell First Than Spectrum
Number analyzed (Participants) | 19 | 26
score on a scale
  "Describe the Sanitizer Quality" Ranging from 0 (thin watery) to 100 (thick, foamy) for Spectrum | 53.21 (19.44) | 39.62 (26.45)
  "Describe the Sanitizer Quality" Ranging from 0 (thin watery) to 100 (thick, foamy) for Purell | 61.21 (26.78) | 49.73 (23.61)
  Sanitizer spread evenly over hands for full coverage (strongly disagree to strongly agree) Spectrum | 84.58 (14.87) | 73.35 (22.00)
  Sanitizer spread evenly over hands for full coverage (strongly disagree to strongly agree) Purell | 82.53 (16.27) | 82.38 (14.34)
  After applying, my hands felt hydrated/moisturized strongly disagree to strongly agree Spectrum | 60.05 (23.28) | 60.85 (22.84)
  After applying, my hands felt hydrated/moisturized strongly disagree to strongly agree Purell | 60.42 (20.86) | 68.58 (19.55)
  Rate the Pleasantness of the Fragrance" (strongly disagree to strongly agree) Spectrum | 0.37 (0.49) | 0.38 (0.50)
  Rate the Pleasantness of the Fragrance" (strongly disagree to strongly agree) Purell | 0.74 (0.45) | 0.73 (0.45)

2. Primary Outcome: Primary Objective Foam Sanitizer User Preference
Description: Healthcare workers' assessment of foam product preference via questionnaire, this was asked "and this question was asked after both *products* had been applied and washed off"
Time Frame: up to 30 mins to complete on a single day; Directly after both products had been applied and washed off.
Population: this question was asked after both products had been applied and washed off
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Spectrum First Then Purell: Arm A participants applied Spectrum hand sanitizer, followed by a washout period, followed by Purell hand sanitizer -question asked after Purell
- Arm B: Purell First Then Spectrum: Arm B participants applied Purell hand sanitizer first, followed by a washout period, followed by applying Spectrum hand sanitizer - question asked after spectrum
Arm/Group | Arm A: Spectrum First Then Purell | Arm B: Purell First Then Spectrum
Number analyzed (Participants) | 19 | 26
Participants
  Spectrum | 4 | 12
  Purell | 15 | 14

3. Primary Outcome: Primary Objective Foam Sanitizer User Preference 2
Description: Participants were asked "If the other product was chosen by the facility, I would object". this was asked in the time window after both products had already been applied and washed off and therefore this question has a different arms grouping than the first set of questions. It was not asked when a given product was on the skin. The participants were blinded to the product being tested at a given time -- so there was no intent to connect this question to the product testing. The facility had clearly labeled wall units with hand sanitizer and all nurses were aware of what brand of product hand sanitizer the facility used.
Time Frame: up to 30 mins to complete on a single day; Directly after both products had been applied and washed off.
Population: Both Arm participants answered the survey question if they would object if their facility switched hand sanitzers from the current product being used at their facility (yes or no). this was asked in the time window after both products had already been applied and washed off and therefore this question has a different arms grouping than the first set of questions. It was not asked when a given product was on the skin.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Spectrum First Then Purell: Arm A participants applied spectrum hand sanitizer first, followed by a washout, followed by applying Purell hand sanitizer
- Arm B: Purell First Than Spectrum: Arm B: participants applied purell hand sanitizer, followed by a washout, then they applied spectrum hand sanitizer.
Arm/Group | Arm A: Spectrum First Then Purell | Arm B: Purell First Than Spectrum
Number analyzed (Participants) | 19 | 26
Participants
  No | 17 | 23
  Yes | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the study duration of 30 mins
Description: No adverse events of any level were noted. These products were already being used regularly by these healthcare professionals in the facility.
Groups:
- Arm A: Spectrum First Then Purell While Using Spectrum: Arm A applied spectrum hand sanitizer first, followed by a washout period, then applied purell hand sanitizer.
  These results report adverse events for group A while using spectrum
- Arm B: Purell First Then Spectrum While Using Purell: Arm B applied Purell hand sanitizer first, followed by a washout period, then applied spectrum hand sanitizer
  These results report adverse events for group B while usuing Purell
- Arm B: Purell First Then Spectrum While Using Spectrum: Arm B applied Purell hand sanitizer first, followed by a washout period, then applied spectrum hand sanitizer
  These results report adverse events for group B while using Spectrum
- Arm A Applied Spectrum Hand Sanitizer Firs Then Purell While Using Purell: Arm A applied spectrum hand sanitizer first, followed by a washout period, then applied purell hand sanitizer.
  These results report adverse events for group A while using Purell
Arm/Group | Arm A: Spectrum First Then Purell While Using Spectrum | Arm B: Purell First Then Spectrum While Using Purell | Arm B: Purell First Then Spectrum While Using Spectrum | Arm A Applied Spectrum Hand Sanitizer Firs Then Purell While Using Purell
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/26 | 0/26 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/26 | 0/26 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/26 | 0/26 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT05755282/Prot_SAP_000.pdf